CLINICAL TRIAL: NCT00396344
Title: The Effect of Glucocorticoid Pre-Treatment on the Systemic Cytokine Response to Endotoxin in Human Volunteers
Brief Title: Cortisol Control of Human Inflammatory Responses to Endotoxin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: CPHS#20361; NIH#AIO51547
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Sepsis
Keywords: Systemic sepsis
MeSH Terms: conditions — Sepsis; Toxemia | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Placebo Comparator): Saline control
  Interventions: Other: Çontrol
- 2 (Experimental)
  Interventions: Drug: Hydrocortisone
- 3 (Experimental)
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Other: Çontrol — Intravenous saline
  Arms: 1
Drug: Hydrocortisone — Intravenous stress dose of hydrocortisone
  Arms: 2
Drug: Hydrocortisone — Intravenous pharmacologic hydrocortisone
  Arms: 3

SUMMARY:
The purpose of the research is to study a common and dangerous medical condition called 'septic shock' that often occurs in critically ill patients. In order to learn about septic shock in humans, we will administer a substance called 'endotoxin' to participants in this study. Endotoxin causes a temporary period of inflammation in the human body, a brief 'virtual' infection. This is an established method for the investigation of inflammation properties. We are interested in how the natural hormone, cortisol, can affect the human response to endotoxin. We know that when cortisol is given at the same time as endotoxin it can decrease the inflammation that occurs due to endotoxin. In this study we will test whether or not cortisol, when given the day before the endotoxin, will work to change the inflammation that occurs due to endotoxin. In order to test this, two-thirds of the study participants will receive cortisol on the day before they receive the endotoxin and one-third of the study participants will receive a placebo (no medication) before the endotoxin.

ELIGIBILITY:
Inclusion Criteria:

* 18 < age < 55
* Weight > 50 kg
* The participant is healthy, without known or suspected medical illness following routine history and physical examination and is expected to easily tolerate the clinical effects of endotoxin.
* The participant does not take any regularly scheduled medication other than thyroid replacement therapy, birth control pills, or estrogenic hormone replacement therapy.

Exclusion Criteria:

* History of chronic disease of any kind such as diabetes, heart disease, cancer, HIV infection, hypertension, asthma, etc.
* History of chronic medication use other than hormone therapy as above
* History of recent acute illness within 30 days prior to study
* Inability to provide informed consent
* History of recent exposure to drugs known to alter immune function including steroids or recent infection (< 3 months)
* Pregnancy
* History of known risk factors for HIV infection (recent multiple partners, sexually transmitted disease and unprotected sex; intravenous drug use; blood transfusion before 1985)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Plasma cytokine responses to in vivo endotoxin administration | 4 Days

SECONDARY OUTCOMES:
Plasma acute phase protein response | 4 Days
Clinical response | 8 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Yeager, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Yeager MP, Rassias AJ, Pioli PA, Beach ML, Wardwell K, Collins JE, Lee HK, Guyre PM. Pretreatment with stress cortisol enhances the human systemic inflammatory response to bacterial endotoxin. Crit Care Med. 2009 Oct;37(10):2727-32. doi: 10.1097/ccm.0b013e3181a592b3. PMID 19885996